CLINICAL TRIAL: NCT04003610
Title: A Phase 2, Open-Label, Randomized, Multicenter Study to Evaluate the Efficacy and Safety of Pemigatinib Plus Pembrolizumab Versus Pemigatinib Alone Versus Standard of Care as First-Line Treatment for Metastatic or Unresectable Urothelial Carcinoma in Cisplatin-Ineligible Participants Whose Tumors Express FGFR3 Mutation or Rearrangement (FIGHT-205)
Brief Title: Pemigatinib + Pembrolizumab vs Pemigatinib Alone vs Standard of Care for Urothelial Carcinoma (FIGHT-205)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The reason this study was terminated was due to a business decision. There were no safety concerns that contributed to this decision.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 54828-205; 2019-000721-50 (EudraCT Number)
Record Dates: First submitted 2019-06-28; First posted 2019-07-01 (Actual); Results first posted 2022-05-25 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Urothelial Carcinoma; Unresectable Urothelial Carcinoma
Keywords: Urothelial carcinoma; fibroblast growth factor receptor (FGFR) inhibitor; FGFR3 mutation; FGFR3 rearrangement; metastatic; unresectable; cisplatin-ineligible
MeSH Terms: conditions — Carcinoma, Transitional Cell; Acrocephalosyndactylia; Neoplasm Metastasis | interventions — pemigatinib; pembrolizumab; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pemigatinib + Pembrolizumab (Experimental): Combination of pemigatinib (13.5 milligrams [mg] once a day orally) plus pembrolizumab (200 mg every 3 weeks [Q3W] intravenously [IV])
  Interventions: Drug: Pemigatinib; Drug: Pembrolizumab
- Pemigatinib (Experimental): Pemigatinib (13.5 mg once a day orally) alone
  Interventions: Drug: Pemigatinib
- Standard of Care (Active Comparator): Either gemcitabine plus carboplatin or pembrolizumab as standard of care. Gemcitabine 1000 mg/meters squared (m^2) IV over 30 minutes on Days 1 and 8, followed by carboplatin (dosed to target area under the concentration-time curve [AUC] of 5 mg/milliliters [mL]/minute [min] or 4.5 mg/mL/min if required per local guidelines) on Day 1 or 2 of each 3-week cycle. Pembrolizumab 200 mg IV on Day 1 of each 21-day treatment cycle for up to 35 cycles or disease progression.
  Interventions: Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Pemigatinib — 13.5 mg once a day orally
  Other Names: INCB054828
  Arms: Pemigatinib; Pemigatinib + Pembrolizumab
Drug: Pembrolizumab — 200 mg Q3W intravenously
  Other Names: Keytruda®
  Arms: Pemigatinib + Pembrolizumab
Drug: Gemcitabine — 1000 mg/m^2 IV over 30 minutes on Days 1 and 8 of each 3-week cycle
  Arms: Standard of Care
Drug: Carboplatin — Dosed to target AUC of 5 mg/mL/min or 4.5 mg/mL/min if required per local guidelines on Day 1 or 2 of each 3-week cycle
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of pemigatinib plus pembrolizumab or pemigatinib alone versus the standard of care for participants with metastatic or unresectable urothelial carcinoma who are not eligible to receive cisplatin, are harboring FGFR3 mutation or rearrangement, and who have not received prior treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented metastatic or unresectable urothelial carcinoma. Both transitional cell and mixed transitional cell histologies are allowed, provided urothelial component is ≥ 50%.
* At least 1 measurable target lesion per RECIST v1.1.
* Must be ineligible to receive cisplatin. Patients ineligible for any platinum-based chemotherapy are allowed.
* Known FGFR3 mutation or rearrangement confirmed by the central laboratory prior to randomization.
* Central laboratory test result of PD-L1 status is mandatory at screening.
* Have received no prior systemic chemotherapy for metastatic or unresectable urothelial carcinoma (except adjuvant platinum-based chemotherapy following radical cystectomy, with recurrence > 12 months from completion of therapy, or neo-adjuvant platinum-based chemotherapy, with recurrence > 12 months since completion of therapy).
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Prior receipt of a selective FGFR inhibitor for any indication or reason.
* Prior receipt of an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent, or with an agent directed to another co-inhibitory T-cell receptor.
* Receipt of anticancer medications or investigational drugs for unresectable and/or metastatic disease.
* Concurrent anticancer therapy, except for treatment allowed per protocol.
* Has disease that is suitable for local therapy administered with curative intent.
* Has tumor with any neuroendocrine or small cell component.
* Current evidence of clinically significant corneal or retinal disorder as confirmed by ophthalmologic examination.
* Has received prior radiotherapy to a metastatic site without the use of chemotherapy radiosensitization within 3 weeks of the first dose of study treatment, with the exception of palliative radiotherapy to bone lesions, which is allowed if completed 2 weeks before the start of study treatment.
* Has central nervous system metastases, unless the participant has completed local therapy (eg, whole brain radiation therapy, surgery, radiosurgery) and has discontinued use of corticosteroids for this indication for at least 4 weeks before starting treatment in this study.
* Known additional malignancy that is progressing or required active treatment within the past 3 years
* Laboratory values outside the protocol-defined range at screening.
* Clinically significant or uncontrolled cardiac disease.
* History of autoimmune disease that has required systemic treatment in past 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2021-04-18 (Actual); Study Completion 2021-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Feliz Vinas, MD, Study Director — Incyte Corporation
Locations (79):
- United States (13):
  - Marin Cancer Care, Greenbrae, California
  - Christiana Care Helen F. Graham Cancer Center, Newark, Delaware
  - Cotton-O'Neil Clinical Research Center, Hematology & Oncology, Marietta, Georgia
  - Simmons Cancer Institute At Siu, Springfield, Illinois
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Smhc Cancer Blood Disorders, Biddeford, Maine
  - Summit Medical Group, Florham Park, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - The Center For Cancer and Blood Disorders, Fort Worth, Texas
  - Onc Consultants Pharmacy 2, Houston, Texas
- Wilhelminenspital, Vienna, Austria
- Belgium (2):
  - Grand Hopital de Charleroi, Charleroi
  - Universitaire Ziekenhuis Leuven - Gasthuisberg, Leuven
- Moncton Hospital - Horizon Health Network, Moncton, New Brunswick, Canada
- Finland (3):
  - Helsinki University Meilahti Tower Hospital, Helsinki
  - Fonk Onkologian Klinikka, Tampere
  - Turku University Hospital, Sct Unit, Turku
- France (10):
  - Centre Hospitalier Universitaire de Besancon, Besançon
  - Groupe Hospitalier Pellegrin Tripode, Bordeaux
  - Polyclinique de Blois, La Chaussée-Saint-Victor
  - Chu Nimes, Nîmes
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - Hopital Cochin Cancerologie, Paris
  - Hopital Europeen Georges Pompidou (Hegp), Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Chu de Strasbourg Hopitaux Universitaires Service D Hematologie, Strasbourg
  - Institut Claudius Regaud Oncopole Toulouse, Toulouse
- Kliniken Maria Hilf, Mönchengladbach, Germany
- University Hospital Waterford, Waterford, Ireland
- Italy (11):
  - Iov - Istituto Oncologico Veneto Irccs, Bari
  - Istituto Tumori Giovanni Paolo Ii Irccs Ospedale Oncologico Bari, Bari
  - L AZIENDA OSPEDALIERO-UNIVERSITARIA DI BOLOGNA POLICLINICO S. ORSOLA ï¿½ MALPIGHI, Bologna
  - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori, Meldola
  - Fondazione Irccs Ca Granda Ospedale Maggiore, Milan
  - Fondazione Irccs Istituto Nazionale Dei Tumori, Milan
  - Ieo Istituto Europeo Di Oncologia Irccs, Milan
  - Istituto Nazionale Tumori Fondazione Irccs G. Pascale, Napoli
  - UNIVERSITï¿½ CAMPUS BIO-MEDICO DI ROMA, Roma
  - Irrcs Instituto Clinico Humanitas, Rozzano
  - Azosp S.Maria Sc Oncologia, Terni
- Japan (21):
  - Chiba University Hospital, Chiba
  - Chiba Cancer Center, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Saitama Medical University International Medical Center, Hidaka-shi
  - Hirosaki University Hospital, Hirosaki-shi
  - Hakodate Goryokaku Hospital, Hokkaido
  - Sapporo Medical University Hospital, Hokkaido
  - Nihon University Itabashi Hospital, Itabashi-ku
  - Nara Medical University Hospital, Kashihara-shi
  - St. Marianna University School of Medicine Hospital, Kawasaki-shi
  - Kagawa University Hospital, Kita-gun
  - Nho Shikoku Cancer Center, Matsuyama
  - Toranomon Hospital, Minatoku
  - Osaka International Cancer Institute, Osaka
  - Saitama Medical Center Jichi Medical University, Saitama-shi
  - Tohoku University Hospital, Sendai
  - Jichi Medical University Hospital, Shimotsuke-shi
  - Keio University Hospital, Shinjuku-ku
  - Osaka University Hospital, Suita-shi
  - National Cancer Center Hospital, Tokyo
  - Toyama University Hospital, Toyama
- Olsztynski Osrodek Onkologiczny Kopernik, Olsztyn, Poland
- Champalimaud Foundation - Champalimaud Centre For the Unknown (Champalimaud Cancer Center), Lisbon, Portugal
- Spitalul Clinic Judetean de Urgenta 'Sf Apostol Andrei' Constanta, Constanța, Romania
- Fakultna Nemocnica S Poliklinikou Zilina, Žilina, Slovakia
- Spain (10):
  - Hospital Clinic I Provincial, Barcelona
  - Ico Institut Catala D Oncologia, Barcelona
  - Ico Girona, Girona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de La Paz, Madrid
  - Hospital Universitario Hm Sanchinarro, Madrid
  - Hospital Puerta de Hierro, Majadahonda
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Barts Health Nhs Trust - St Bartholomews Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted (enrolled participants) at 7 sites located in France, Italy, Spain, and Japan.
Groups:
- Pemigatinib 13.5 mg: Pemigatinib was self-administered at 13.5 milligrams (mg) once daily (QD) orally (PO) until disease progression during each 21-day treatment cycle. Participants not reaching the target serum phosphate level (> 5.5 mg/deciliter [dL]) during Cycle 1 despite being study drug compliant increased the daily pemigatinib dose to 18 mg starting at Cycle 2 as long as they were not experiencing an ongoing Grade 2 or higher treatment-related adverse event (AE).
- Pemigatinib 13.5 mg Plus Pembrolizumab 200 mg: Pemigatinib was self-administered at 13.5 mg QD PO until disease progression during each 21-day treatment cycle. Participants not reaching the target serum phosphate level (> 5.5 mg/dL) during Cycle 1 despite being study drug compliant increased the daily pemigatinib dose to 18 mg starting at Cycle 2 as long as they were not experiencing an ongoing Grade 2 or higher treatment-related AE. Pembrolizumab 200 mg was administered intravenously (IV) on Day 1 of each 21-day treatment cycle for up to 35 cycles or disease progression.
- Gemcitabine 1000 mg/m^2 Plus Carboplatin or Pembrolizumab 200 mg: Participants received either gemcitabine plus carboplatin or pembrolizumab as standard of care. Participants received gemcitabine 1000 mg/meters squared (m^2) IV over 30 minutes on Days 1 and 8 of each 3-week treatment cycle, followed by carboplatin (dosed to target area under the concentration-time curve [AUC] of 5 mg/milliliters [mL]/minute [min] or 4.5 mg/mL/min if required per local guidelines) on Day 1 or Day 2 of each 3-week treatment cycle. Treatment continued for 4 to 6 cycles (or per institutional standards) until disease progression or intolerable toxicity. Pembrolizumab 200 mg was administered IV on Day 1 of each 21-day treatment cycle for up to 35 cycles or disease progression.
Period: Overall Study
Arm/Group | Pemigatinib 13.5 mg | Pemigatinib 13.5 mg Plus Pembrolizumab 200 mg | Gemcitabine 1000 mg/m^2 Plus Carboplatin or Pembrolizumab 200 mg
Started | 0 | 1 | 6
Completed | 0 | 0 | 0
Not Completed | 0 | 1 | 6
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Death | 0 | 0 | 3
Not completed — Study Terminated by Sponsor | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in the pemigatinib 13.5 mg treatment arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemigatinib 13.5 mg | Pemigatinib 13.5 mg Plus Pembrolizumab 200 mg | Gemcitabine 1000 mg/m^2 Plus Carboplatin or Pembrolizumab 200 mg | Total
Number analyzed (Participants) | 0 | 1 | 6 | 7
Age, Customized [Count of Participants; unit: Participants]
  57 to 84 years old | 0 | 1 | 6 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 4 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male |  | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 2 | NA — Total not calculated because data are not available (NA) in one or more arms.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Not Hispanic or Latino |  | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 5 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported |  | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 1 | NA — Total not calculated because data are not available (NA) in one or more arms.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian |  | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 3 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian or Other Pacific Islander |  | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American |  | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  White |  | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 3 | NA — Total not calculated because data are not available (NA) in one or more arms.
  More than one race |  | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported |  | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the randomization date until the date of disease progression (as measured by a blinded independent central review [BICR] per Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST v1.1]) or death due to any cause, whichever occurred first.
Time Frame: up to 130 days
Population: Intent-to-Treat (ITT) Population: all participants who were randomized into the study. Treatment groups for this population were to be determined according to the treatment assignment at the time of randomization. The 95% confidence intervals were calculated using the Brookmeyer and Crowley's method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemigatinib 13.5 mg | Pemigatinib 13.5 mg Plus Pembrolizumab 200 mg | Gemcitabine 1000 mg/m^2 Plus Carboplatin or Pembrolizumab 200 mg
Number analyzed (Participants) | 0 | 1 | 6
months |  | 1.81 [NA to NA] — The upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. | 2.12 [1.51 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died.

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until death due to any cause.
Time Frame: up to 225 days
Population: ITT Population. The 95% confidence intervals were calculated using the Brookmeyer and Crowley's method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemigatinib 13.5 mg | Pemigatinib 13.5 mg Plus Pembrolizumab 200 mg | Gemcitabine 1000 mg/m^2 Plus Carboplatin or Pembrolizumab 200 mg
Number analyzed (Participants) | 0 | 1 | 6
months |  | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants died. | NA [1.51 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants died.

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the proportion of participants with a best overall response of complete response (CR) or partial response (PR) per RECIST v1.1 (as measured by BICR).
Time Frame: up to 148 days
Population: Intent-to-Treat (ITT) Population: all participants who were randomized into the study. Treatment groups for this population were to be determined according to the treatment assignment at the time of randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Pemigatinib 13.5 mg | Pemigatinib 13.5 mg Plus Pembrolizumab 200 mg | Gemcitabine 1000 mg/m^2 Plus Carboplatin or Pembrolizumab 200 mg
Number analyzed (Participants) | 0 | 1 | 6
percentage of participants |  | 0 | 0

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the date of the first assessment of CR or PR until the date of the first disease progression (per RECIST v1.1) or death, whichever occurred first (as measured by BICR).
Time Frame: up to 148 days
Population: As measured by BICR, there were no responders; thus, DOR was not calculated.
Arm/Group | Pemigatinib 13.5 mg | Pemigatinib 13.5 mg Plus Pembrolizumab 200 mg | Gemcitabine 1000 mg/m^2 Plus Carboplatin or Pembrolizumab 200 mg
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: A treatment-emergent adverse event was defined as an adverse event that was either reported for the first time or the worsening of a pre-existing event after the first dose of study drug until 30 days after the last dose of study drug.
Time Frame: up to 178 days
Population: Safety Population: all randomized participants who received at least one dose of study treatment. Treatment groups for this population were to be determined according to the actual treatment the participant received regardless of assigned study drug treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pemigatinib 13.5 mg | Pemigatinib 13.5 mg Plus Pembrolizumab 200 mg | Gemcitabine 1000 mg/m^2 Plus Carboplatin or Pembrolizumab 200 mg
Number analyzed (Participants) | 0 | 1 | 6
Participants |  | 1 | 6

6. Secondary Outcome: EORTC QLQ-C30 Score
Description: The European Organization for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) contains 30 items and measures 5 functional dimensions (i.e., physical, role, emotional, cognitive, and social), 3 symptom items (i.e., fatigue, nausea/vomiting, and pain), 6 single items (i.e., dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and financial impact), and a global health and quality of life scale. For each scale and single item, a linear transformation was applied to standardize the scores between 0 (worst) and 100 (best) as described in the EORTC QLQ-C30 Scoring Manual.
Time Frame: up to 160 days
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Gemcitabine 1000 mg/m^2 Plus carboplatinGemcitabine 1000 mg/m^2 Plus Carboplatin: Participants received either gemcitabine plus carboplatin or pembrolizumab as standard of care. Participants received gemcitabine 1000 mg/meters squared (m^2) IV over 30 minutes on Days 1 and 8 of each 3-week treatment cycle, followed by carboplatin (dosed to target area under the concentration-time curve [AUC] of 5 mg/milliliters [mL]/minute [min] or 4.5 mg/mL/min if required per local guidelines) on Day 1 or Day 2 of each 3-week treatment cycle. Treatment continued for 4 to 6 cycles (or per institutional standards) until disease progression or intolerable toxicity. Pembrolizumab 200 mg was administered IV on Day 1 of each 21-day treatment cycle for up to 35 cycles or disease progression.
Arm/Group | Pemigatinib 13.5 mg | Pemigatinib 13.5 mg Plus Pembrolizumab 200 mg | Gemcitabine 1000 mg/m^2 Plus carboplatinGemcitabine 1000 mg/m^2 Plus Carboplatin
Number analyzed (Participants) | 0 | 1 | 5
scores on a scale
  Appetite Loss, Baseline |  | 33.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis. | 26.7 (36.51)
  Appetite Loss, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Appetite Loss, Cycle 3 Day 1 |  |  | 16.7 (23.57)
  Appetite Loss, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Appetite Loss, Cycle 6 Day 1 |  |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Appetite Loss, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Appetite Loss, Follow Up |  |  | 66.7 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Cognitive Functioning, Baseline |  | 66.7 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis. | 66.7 (20.41)
  Cognitive Functioning, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Cognitive Functioning, Cycle 3 Day 1 |  |  | 91.7 (11.79)
  Cognitive Functioning, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Cognitive Functioning, Cycle 6 Day 1 |  |  | 66.7 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Cognitive Functioning, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Cognitive Functioning, Follow Up |  |  | 83.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Constipation, Baseline |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis. | 40.0 (27.89)
  Constipation, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Constipation, Cycle 3 Day 1 |  |  | 16.7 (23.57)
  Constipation, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Constipation, Cycle 6 Day 1 |  |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Constipation, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Constipation, Follow Up |  |  | 33.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Diarrhea, Baseline |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis. | 20.0 (44.72)
  Diarrhea, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Diarrhea, Cycle 3 Day 1 |  |  | 0.0 (0.0)
  Diarrhea, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Diarrhea, Cycle 6 Day 1 |  |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Diarrhea, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Diarrhea, Follow Up |  |  | 33.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Dyspnea, Baseline |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis. | 26.7 (27.89)
  Dyspnea, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Dyspnea, Cycle 3 Day 1 |  |  | 16.7 (23.57)
  Dyspnea, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Dyspnea, Cycle 6 Day 1 |  |  | 33.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Dyspnea, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Dyspnea, Follow Up |  |  | 66.7 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Emotional Functioning, Baseline |  | 50.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis. | 73.3 (19.00)
  Emotional Functioning, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Emotional Functioning, Cycle 3 Day 1 |  |  | 87.5 (5.89)
  Emotional Functioning, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Emotional Functioning, Cycle 6 Day 1 |  |  | 91.7 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Emotional Functioning, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Emotional Functioning, Follow Up |  |  | 100.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Fatigue, Baseline |  | 44.4 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis. | 46.7 (36.35)
  Fatigue, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Fatigue, Cycle 3 Day 1 |  |  | 50.0 (39.28)
  Fatigue, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Fatigue, Cycle 6 Day 1 |  |  | 33.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Fatigue, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Fatigue, Follow Up |  |  | 55.6 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Financial Difficulties, Baseline |  | 33.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis. | 20.0 (18.26)
  Financial Difficulties, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Financial Difficulties, Cycle 3 Day 1 |  |  | 16.7 (23.57)
  Financial Difficulties, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Financial Difficulties, Cycle 6 Day 1 |  |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Financial Difficulties, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Financial Difficulties, Follow Up |  |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Global Health Status/Quality of Life (QoL), Baseline |  | 16.7 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis. | 51.7 (31.95)
  Global Health Status/QoL, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Global Health Status/QoL, Cycle 3 Day 1 |  |  | 66.7 (11.79)
  Global Health Status/QoL, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Global Health Status/QoL, Cycle 6 Day 1 |  |  | 66.7 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Global Health Status/QoL, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Global Health Status/QoL, Follow Up |  |  | 50.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Insomnia, Baseline |  | 33.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis. | 46.7 (38.01)
  Insomnia, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Insomnia, Cycle 3 Day 1 |  |  | 33.3 (47.14)
  Insomnia, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Insomnia, Cycle 6 Day 1 |  |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Insomnia, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Insomnia, Follow Up |  |  | 66.7 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Nausea and Vomiting, Baseline |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis. | 6.7 (9.13)
  Nausea and Vomiting, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Nausea and Vomiting, Cycle 3 Day 1 |  |  | 8.3 (11.79)
  Nausea and Vomiting, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Nausea and Vomiting, Cycle 6 Day 1 |  |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Nausea and Vomiting, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Nausea and Vomiting, Follow Up |  |  | 16.7 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Pain, Baseline |  | 50.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis. | 40.0 (43.46)
  Pain, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Pain, Cycle 3 Day 1 |  |  | 41.7 (11.79)
  Pain, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Pain, Cycle 6 Day 1 |  |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Pain, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Pain, Follow Up |  |  | 16.7 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Physical Functioning, Baseline |  | 73.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis. | 65.3 (26.83)
  Physical Functioning, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Physical Functioning, Cycle 3 Day 1 |  |  | 33.3 (47.14)
  Physical Functioning, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Physical Functioning, Cycle 6 Day 1 |  |  | 66.7 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Physical Functioning, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Physical Functioning, Follow Up |  |  | 40.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Role Functioning, Baseline |  | 66.7 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis. | 56.7 (40.14)
  Role Functioning, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Role Functioning, Cycle 3 Day 1 |  |  | 33.3 (47.14)
  Role Functioning, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Role Functioning, Cycle 6 Day 1 |  |  | 66.7 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Role Functioning, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Role Functioning, Follow Up |  |  | 33.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Social Functioning, Baseline |  | 66.7 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis. | 53.3 (36.13)
  Social Functioning, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Social Functioning, Cycle 3 Day 1 |  |  | 66.7 (0.00)
  Social Functioning, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Social Functioning, Cycle 6 Day 1 |  |  | 66.7 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Social Functioning, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Social Functioning, Follow Up |  |  | 83.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.

7. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Score
Description: The European Organization for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) contains 30 items and measures 5 functional dimensions (i.e., physical, role, emotional, cognitive, and social), 3 symptom items (i.e., fatigue, nausea/vomiting, and pain), 6 single items (i.e., dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and financial impact), and a global health and quality of life scale. For each scale and single item, a linear transformation was applied to standardize the scores between 0 (worst) and 100 (best) as described in the EORTC QLQ-C30 Scoring Manual. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; up to 160 days
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pemigatinib 13.5 mg | Pemigatinib 13.5 mg Plus Pembrolizumab 200 mg | Gemcitabine 1000 mg/m^2 Plus Carboplatin or Pembrolizumab 200 mg
Number analyzed (Participants) | 0 | 1 | 5
scores on a scale
  Appetite Loss, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Appetite Loss, Cycle 3 Day 1 |  |  | -16.7 (23.57)
  Appetite Loss, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Appetite Loss, Cycle 6 Day 1 |  |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Appetite Loss, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Appetite Loss, Follow Up |  |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Cognitive Functioning, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Cognitive Functioning, Cycle 3 Day 1 |  |  | 33.3 (23.57)
  Cognitive Functioning, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Cognitive Functioning, Cycle 6 Day 1 |  |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Cognitive Functioning, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Cognitive Functioning, Follow Up |  |  | 33.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Constipation, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Constipation, Cycle 3 Day 1 |  |  | -33.3 (0.00)
  Constipation, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Constipation, Cycle 6 Day 1 |  |  | -33.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Constipation, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Constipation, Follow Up |  |  | -33.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Diarrhea, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Diarrhea, Cycle 3 Day 1 |  |  | -50.0 (70.71)
  Diarrhea, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Diarrhea, Cycle 6 Day 1 |  |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Diarrhea, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Diarrhea, Follow Up |  |  | -66.7 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Dyspnea, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Dyspnea, Cycle 3 Day 1 |  |  | 0.0 (0.00)
  Dyspnea, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Dyspnea, Cycle 6 Day 1 |  |  | 33.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Dyspnea, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Dyspnea, Follow Up |  |  | 33.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Emotional Functioning, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Emotional Functioning, Cycle 3 Day 1 |  |  | 12.5 (29.46)
  Emotional Functioning, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Emotional Functioning, Cycle 6 Day 1 |  |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Emotional Functioning, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Emotional Functioning, Follow Up |  |  | 41.7 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Fatigue, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Fatigue, Cycle 3 Day 1 |  |  | -11.1 (15.71)
  Fatigue, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Fatigue, Cycle 6 Day 1 |  |  | 11.1 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Fatigue, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Fatigue, Follow Up |  |  | -44.4 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Financial Difficulties, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Financial Difficulties, Cycle 3 Day 1 |  |  | 0.0 (0.00)
  Financial Difficulties, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Financial Difficulties, Cycle 6 Day 1 |  |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Financial Difficulties, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Financial Difficulties, Follow Up |  |  | -33.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Global Health Status/QoL, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Global Health Status/QoL, Cycle 3 Day 1 |  |  | 33.3 (35.36)
  Global Health Status/QoL, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Global Health Status/QoL, Cycle 6 Day 1 |  |  | 16.7 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Global Health Status/QoL, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Global Health Status/QoL, Follow Up |  |  | 33.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Insomnia, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Insomnia, Cycle 3 Day 1 |  |  | -16.7 (23.57)
  Insomnia, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Insomnia, Cycle 6 Day 1 |  |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Insomnia, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Insomnia, Follow Up |  |  | -33.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Nausea and Vomiting, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Nausea and Vomiting, Cycle 3 Day 1 |  |  | 0.0 (0.00)
  Nausea and Vomiting, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Nausea and Vomiting, Cycle 6 Day 1 |  |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Nausea and Vomiting, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Nausea and Vomiting, Follow Up |  |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Pain, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Pain, Cycle 3 Day 1 |  |  | -8.3 (58.93)
  Pain, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Pain, Cycle 6 Day 1 |  |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Pain, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Pain, Follow Up |  |  | -83.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Physical Functioning, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Physical Functioning, Cycle 3 Day 1 |  |  | -26.7 (37.71)
  Physical Functioning, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Physical Functioning, Cycle 6 Day 1 |  |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Physical Functioning, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Physical Functioning, Follow Up |  |  | -13.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Role Functioning, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Role Functioning, Cycle 3 Day 1 |  |  | 0.0 (0.00)
  Role Functioning, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Role Functioning, Cycle 6 Day 1 |  |  | 0.0 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Role Functioning, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Role Functioning, Follow Up |  |  | 33.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Social Functioning, Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 2
  Social Functioning, Cycle 3 Day 1 |  |  | 41.7 (11.79)
  Social Functioning, Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Social Functioning, Cycle 6 Day 1 |  |  | 33.3 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Social Functioning, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Social Functioning, Follow Up |  |  | 66.7 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.

8. Secondary Outcome: Number of Participants With the Indicated EQ-5D-5L Dimension Scores
Description: The EQ-5D-5L is a standardized instrument for use as a measure of health outcome. The EQ-5D-5L descriptive system is composed of 5 dimensions (mobility, self-case, usual activities, pain/discomfort, and anxiety/depression). Each dimension has 5 response levels, which are coded by single-digit numbers: 1 = no problems, 2 = slight problems, 3 = moderate problems, 4 = severe problems, 5 = unable to/extreme problems. The EQ-5D-5L also includes a graded (0 [worst overall health] to 100 [best overall health]) vertical visual analog scale that provides a quantitative measure of the participant's perception of their overall health.
Time Frame: up to 160 days
Population: ITT Population. Only participants with available data were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Pemigatinib 13.5 mg | Pemigatinib 13.5 mg Plus Pembrolizumab 200 mg | Gemcitabine 1000 mg/m^2 Plus Carboplatin or Pembrolizumab 200 mg
Number analyzed (Participants) | 0 | 1 | 5
Participants
  Anxiety/Depression, Baseline: 1 |  | 0 | 3
  Anxiety/Depression, Baseline: 2 |  | 0 | 0
  Anxiety/Depression, Baseline: 3 |  | 1 | 1
  Anxiety/Depression, Baseline: 4 |  | 0 | 1
  Anxiety/Depression, Baseline: 5 |  | 0 | 0
  Anxiety/Depression, Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Anxiety/Depression, Cycle 4 Day 1: 1 |  |  | 1
  Anxiety/Depression, Cycle 4 Day 1: 2 |  |  | 0
  Anxiety/Depression, Cycle 4 Day 1: 3 |  |  | 0
  Anxiety/Depression, Cycle 4 Day 1: 4 |  |  | 0
  Anxiety/Depression, Cycle 4 Day 1: 5 |  |  | 0
  Anxiety/Depression, Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Anxiety/Depression, Cycle 7 Day 1: 1 |  |  | 1
  Anxiety/Depression, Cycle 7 Day 1: 2 |  |  | 0
  Anxiety/Depression, Cycle 7 Day 1: 3 |  |  | 0
  Anxiety/Depression, Cycle 7 Day 1: 4 |  |  | 0
  Anxiety/Depression, Cycle 7 Day 1: 5 |  |  | 0
  Anxiety/Depression, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Anxiety/Depression, Follow Up: 1 |  |  | 1
  Anxiety/Depression, Follow Up: 2 |  |  | 0
  Anxiety/Depression, Follow Up: 3 |  |  | 0
  Anxiety/Depression, Follow Up: 4 |  |  | 0
  Anxiety/Depression, Follow Up: 5 |  |  | 0
  Mobility, Baseline: 1 |  | 0 | 1
  Mobility, Baseline: 2 |  | 0 | 2
  Mobility, Baseline: 3 |  | 1 | 2
  Mobility, Baseline: 4 |  | 0 | 0
  Mobility, Baseline: 5 |  | 0 | 0
  Mobility, Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Mobility, Cycle 4 Day 1: 1 |  |  | 0
  Mobility, Cycle 4 Day 1: 2 |  |  | 1
  Mobility, Cycle 4 Day 1: 3 |  |  | 0
  Mobility, Cycle 4 Day 1: 4 |  |  | 0
  Mobility, Cycle 4 Day 1: 5 |  |  | 0
  Mobility, Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Mobility, Cycle 7 Day 1: 1 |  |  | 0
  Mobility, Cycle 7 Day 1: 2 |  |  | 1
  Mobility, Cycle 7 Day 1: 3 |  |  | 0
  Mobility, Cycle 7 Day 1: 4 |  |  | 0
  Mobility, Cycle 7 Day 1: 5 |  |  | 0
  Mobility, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Mobility, Follow Up: 1 |  |  | 0
  Mobility, Follow Up: 2 |  |  | 0
  Mobility, Follow Up: 3 |  |  | 0
  Mobility, Follow Up: 4 |  |  | 0
  Mobility, Follow Up: 5 |  |  | 1
  Pain/Discomfort, Baseline: 1 |  | 0 | 2
  Pain/Discomfort, Baseline: 2 |  | 0 | 1
  Pain/Discomfort, Baseline: 3 |  | 1 | 0
  Pain/Discomfort, Baseline: 4 |  | 0 | 2
  Pain/Discomfort, Baseline: 5 |  | 0 | 0
  Pain/Discomfort, Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Pain/Discomfort, Cycle 4 Day 1: 1 |  |  | 1
  Pain/Discomfort, Cycle 4 Day 1: 2 |  |  | 0
  Pain/Discomfort, Cycle 4 Day 1: 3 |  |  | 0
  Pain/Discomfort, Cycle 4 Day 1: 4 |  |  | 0
  Pain/Discomfort, Cycle 4 Day 1: 5 |  |  | 0
  Pain/Discomfort, Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Pain/Discomfort, Cycle 7 Day 1: 1 |  |  | 0
  Pain/Discomfort, Cycle 7 Day 1: 2 |  |  | 0
  Pain/Discomfort, Cycle 7 Day 1: 3 |  |  | 1
  Pain/Discomfort, Cycle 7 Day 1: 4 |  |  | 0
  Pain/Discomfort, Cycle 7 Day 1: 5 |  |  | 0
  Pain/Discomfort, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Pain/Discomfort, Follow Up: 1 |  |  | 0
  Pain/Discomfort, Follow Up: 2 |  |  | 0
  Pain/Discomfort, Follow Up: 3 |  |  | 1
  Pain/Discomfort, Follow Up: 4 |  |  | 0
  Pain/Discomfort, Follow Up: 5 |  |  | 0
  Self-care, Baseline: 1 |  | 0 | 3
  Self-care, Baseline: 2 |  | 1 | 0
  Self-care, Baseline: 3 |  | 0 | 2
  Self-care, Baseline: 4 |  | 0 | 0
  Self-care, Baseline: 5 |  | 0 | 0
  Self-care, Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Self-care, Cycle 4 Day 1: 1 |  |  | 0
  Self-care, Cycle 4 Day 1: 2 |  |  | 1
  Self-care, Cycle 4 Day 1: 3 |  |  | 0
  Self-care, Cycle 4 Day 1: 4 |  |  | 0
  Self-care, Cycle 4 Day 1: 5 |  |  | 0
  Self-care, Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Self-care, Cycle 7 Day 1: 1 |  |  | 0
  Self-care, Cycle 7 Day 1: 2 |  |  | 1
  Self-care, Cycle 7 Day 1: 3 |  |  | 0
  Self-care, Cycle 7 Day 1: 4 |  |  | 0
  Self-care, Cycle 7 Day 1: 5 |  |  | 0
  Self-care, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Self-care, Follow Up: 1 |  |  | 0
  Self-care, Follow Up: 2 |  |  | 0
  Self-care, Follow Up: 3 |  |  | 1
  Self-care, Follow Up: 4 |  |  | 0
  Self-care, Follow Up: 5 |  |  | 0
  Usual Activities, Baseline: 1 |  | 0 | 2
  Usual Activities, Baseline: 2 |  | 0 | 1
  Usual Activities, Baseline: 3 |  | 1 | 2
  Usual Activities, Baseline: 4 |  | 0 | 0
  Usual Activities, Baseline: 5 |  | 0 | 0
  Usual Activities, Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Usual Activities, Cycle 4 Day 1: 1 |  |  | 0
  Usual Activities, Cycle 4 Day 1: 2 |  |  | 1
  Usual Activities, Cycle 4 Day 1: 3 |  |  | 0
  Usual Activities, Cycle 4 Day 1: 4 |  |  | 0
  Usual Activities, Cycle 4 Day 1: 5 |  |  | 0
  Usual Activities, Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Usual Activities, Cycle 7 Day 1: 1 |  |  | 0
  Usual Activities, Cycle 7 Day 1: 2 |  |  | 1
  Usual Activities, Cycle 7 Day 1: 3 |  |  | 0
  Usual Activities, Cycle 7 Day 1: 4 |  |  | 0
  Usual Activities, Cycle 7 Day 1: 5 |  |  | 0
  Usual Activities, Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Usual Activities, Follow Up: 1 |  |  | 0
  Usual Activities, Follow Up: 2 |  |  | 0
  Usual Activities, Follow Up: 3 |  |  | 0
  Usual Activities, Follow Up: 4 |  |  | 1
  Usual Activities, Follow Up: 5 |  |  | 0

9. Secondary Outcome: Change From Baseline in the EQ-5D-5L EQ Visual Analog Scale Score
Description: as for outcome 8
Time Frame: Baseline; up to 160 days
Population: ITT Population. Only participants with available data were analyzed
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pemigatinib 13.5 mg | Pemigatinib 13.5 mg Plus Pembrolizumab 200 mg | Gemcitabine 1000 mg/m^2 Plus Carboplatin or Pembrolizumab 200 mg
Number analyzed (Participants) | 0 | 1 | 5
scores on a scale
  Baseline |  | 40 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis. | 52 (30.54)
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Cycle 4 Day 1 |  |  | 5 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Cycle 7 Day 1 |  |  | 5 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.
  Follow Up: number analyzed (Participants) | 0 | 0 | 1
  Follow Up |  |  | 30 (NA) — A standard deviation was not calculated when only 1 participant contributed to the analysis.

ADVERSE EVENTS:
Time Frame: up to 178 days. Deaths were monitored for up to 225 days. Treatment-emergent adverse events (TEAEs) were monitored for up to 178 days (for up to 30 days after last dose of study drug).
Description: TEAEs, defined as adverse events that were either reported for the first time or the worsening of pre-existing events after the first dose of study drug until 30 days after the last dose of study drug, are reported for members of the Safety Population (all randomized participants who received at least one dose of study treatment).
Arm/Group | Pemigatinib 13.5 mg | Pemigatinib 13.5 mg Plus Pembrolizumab 200 mg | Gemcitabine 1000 mg/m^2 Plus Carboplatin or Pembrolizumab 200 mg
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1 | 3/6
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/1 | 1/6
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemigatinib 13.5 mg (N=0) | Pemigatinib 13.5 mg Plus Pembrolizumab 200 mg (N=1) | Gemcitabine 1000 mg/m^2 Plus Carboplatin or Pembrolizumab 200 mg (N=6)
Bone pain (Musculoskeletal and connective tissue disorders) | NA | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | NA | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemigatinib 13.5 mg (N=0) | Pemigatinib 13.5 mg Plus Pembrolizumab 200 mg (N=1) | Gemcitabine 1000 mg/m^2 Plus Carboplatin or Pembrolizumab 200 mg (N=6)
Abdominal pain (Gastrointestinal disorders) | NA | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | NA | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | NA | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | NA | 1 (1) | 0 (0)
Asthenia (General disorders) | NA | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | NA | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | NA | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | NA | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | NA | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | NA | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | NA | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | NA | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | NA | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | NA | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | NA | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | NA | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | NA | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | NA | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | NA | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | NA | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | NA | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | NA | 0 (0) | 1 (1)
Hypofibrinogenaemia (Blood and lymphatic system disorders) | NA | 0 (0) | 1 (1)
Malaise (General disorders) | NA | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | NA | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | NA | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | NA | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | NA | 0 (0) | 1 (1)
Penile pain (Reproductive system and breast disorders) | NA | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | NA | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | NA | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | NA | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | NA | 1 (1) | 0 (0)
Vascular pain (Vascular disorders) | NA | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | NA | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The Sponsor made a decision unrelated to safety to halt study enrollment. Due to early termination of the study with only 7 participants, no analysis of efficacy endpoints was done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT04003610/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT04003610/SAP_001.pdf